CLINICAL TRIAL: NCT02417974
Title: Prevention of Recurrence of Crohn's Disease by Fecal Microbiota Therapy (FMT)
Acronym: FMT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low enrollment was exacerbated by a covid policy related study suspension so the research was stopped.
Sponsor: Boston Medical Center (Other)
Collaborators: Brigham and Women's Hospital (Other); Beth Israel Deaconess Medical Center (Other); Massachusetts Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: H-34244
Record Dates: First submitted 2015-04-01; First posted 2015-04-16 (Estimated); Results first posted 2022-03-24 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-02

CONDITIONS: Crohn's Disease
Keywords: Prevention; Recurrence; Fecal Microbiota Therapy
MeSH Terms: conditions — Crohn Disease; Recurrence | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fecal Microbiota Transplant (FMT) (Experimental): Fecal Microbiota Transplant (FMT) via colonoscopy
  Interventions: Biological: Fecal Microbiota Transplant (FMT)
- Control (No Intervention): No Fecal Microbiota Transplant (FMT) via colonoscopy

INTERVENTIONS:
Biological: Fecal Microbiota Transplant (FMT) — Fecal Microbiota Transplant (FMT)
  Other Names: Fecal Transplant; Stool Transplant
  Arms: Fecal Microbiota Transplant (FMT)

SUMMARY:
The objective of this trial is to assess if Fecal Microbiota Therapy (FMT) can reduce the risk of endoscopic recurrence of Crohn's disease (CD) in patients after intestinal resection. The specific outcomes of FMT to be examined are: 1) endoscopic appearance, 2) clinical symptoms, 3) safety and tolerability, and 4) microbial diversity. The research team hypothesizes that FMT will prevent establishment of "pro-inflammatory" microbiome after surgery, leading to a reduced probability of recurrence of macroscopic inflammation. It is also hypothesized that FMT will be safe and well-tolerated in these patients.

ELIGIBILITY:
Inclusion Criteria (Patients):

* Adults (age > 18)
* Confirmed diagnosis of Crohn's disease (CD), based on endoscopy, histology and imaging (confirmed by Study PI for each site)
* Ileo-cecal resection or terminal ileal resection for CD within 30 days prior to enrollment
* Resection margins & anastomosis free of active inflammation based on histology and surgical description (confirmed by Study PI for each site)
* No therapy to prevent post-operative recurrence of CD. A 30-day wash-out period for anti- tumor necrosis factors (TNF)s, thiopurines, antibiotics will be required prior to enrollment.

Exclusion Criteria (Patients):

* Diagnosis of indeterminate colitis
* Women who are pregnant or nursing
* Patients who are unable to give informed consent
* Patients who are unable or unwilling to undergo colonoscopy with moderate sedation (>ASA class II)
* Patients who have previously undergone FMT
* Patients who have a confirmed malignancy or cancer
* Participation in a clinical trial in the preceding 30 days or simultaneously during this trial
* Probiotic use within 30 days of start date
* Decompensated cirrhosis
* Congenital or acquired immunodeficiencies
* Chronic kidney disease as defined by a GFR <60mL/min/1.73m2 44
* History of rheumatic heart disease, endocarditis, or valvular disease due to risk of bacteremia from colonoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2021-02-04 (Actual); Study Completion 2021-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan C Moss, MD PhD, Principal Investigator — Boston Medical Center
Locations (2):
- United States (2):
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fecal Microbiota Transplant (FMT) | Control
Started | 15 | 9
Completed | 15 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fecal Microbiota Transplant (FMT) | Control | Total
Number analyzed (Participants) | 15 | 9 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 39 (7) | 46 (6) | 41 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 16
  Male | 5 | 3 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 9 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 9 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 9 | 24
Prior resection [Count of Participants; unit: Participants] | 0 | 0 | 0
Smoker [Count of Participants; unit: Participants] | 1 | 0 | 1
Montreal B3 classification [Count of Participants; unit: Participants] — Montreal B3 indicates penetrating Crohn's disease.
  Participants | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Endoscopic Recurrence
Description: Percentage of patients in each arm of the trial who develop endoscopic recurrence within 6 months of ileo-cecal resection. "Endoscopic recurrence" will be defined as a Rutgeert's score of greater than i2
Time Frame: within 6 months of ileo-cecal resection
Measure: Number; unit: percentage of participants
Arm/Group | Fecal Microbiota Transplant (FMT) | Control
Number analyzed (Participants) | 15 | 9
percentage of participants | 20 | 0

2. Secondary Outcome: Change in Microbial Diversity: Shannon Diversity Index
Description: The Shannon Diversity Index is a measure of entropy and is a function of the distribution of the total number of organisms across all of the species. If S is the total number of species in the sample and p_i is the number of organisms in the i-th species divided by the total number of organisms, then Diversity = -Σ p_i log(p_i). Lower values indicate more diversity while higher values indicate less diversity.
Time Frame: baseline, 4, 12, and 26 weeks
Population: There was insufficient data collected for any of the timeframes to calculate the Shannon Diversity Index.
Arm/Group | Fecal Microbiota Transplant (FMT) | Control
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Participants in Clinical Remission at 26 Weeks
Description: Clinical remission is defined as having a Harvey Bradshaw Index (HBI) score <5 at week 26. The HBI can range from 0 to 18 and higher scores are associated with more severe disease.
Time Frame: 26 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Fecal Microbiota Transplant (FMT) | Control
Number analyzed (Participants) | 15 | 9
Participants | 14 | 5

4. Secondary Outcome: Adverse Events Frequency
Description: Number of participants with adverse events
Time Frame: 4, 12, and 26 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Fecal Microbiota Transplant (FMT) | Control
Number analyzed (Participants) | 15 | 9
Participants
  4 weeks | 2 | 1
  12 weeks | 0 | 2
  26 weeks | 0 | 3

ADVERSE EVENTS:
Time Frame: 26 weeks
Arm/Group | Fecal Microbiota Transplant (FMT) | Control
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/15 | 1/9
Other Adverse Events (participants affected / at risk) | 11/15 | 6/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fecal Microbiota Transplant (FMT) (N=15) | Control (N=9)
Hospitalization (Gastrointestinal disorders) | 0 (0) | 1 (1) — Ed visit for diarrhea
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fecal Microbiota Transplant (FMT) (N=15) | Control (N=9)
Symptoms (Gastrointestinal disorders) | 11 (11) | 6 (7) — Diarrhea

LIMITATIONS AND CAVEATS:
Low enrollment was exacerbated by a covid policy related study suspension so the research was stopped.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-10): https://cdn.clinicaltrials.gov/large-docs/74/NCT02417974/Prot_SAP_000.pdf